CLINICAL TRIAL: NCT05057650
Title: African American Health and Nutrition Intervention: Help Everyone Assess Risk Today: LEnten Nutrition Study (HEART-LENS) "Giving up Unhealthy Food for Lent"
Brief Title: Help Everyone Assess Risk Today: LEnten Nutrition Study (HEART-LENS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Kim Allan Williams, Chief, Cardiology Division, James B. Herrick Professor of Medicine, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19020103
Record Dates: First submitted 2021-08-09; First posted 2021-09-27 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Morbidity; Risk Reduction; Nutrition Disorders
Keywords: Nutrition Intervention; plant-based nutrition; cardiovascular risk modification
MeSH Terms: conditions — Risk Reduction Behavior; Nutrition Disorders | interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Vegan food for 5 weeks: approximately 50 participants volunteered for the intervention.
  Interventions: Dietary Supplement: Vegan diet

INTERVENTIONS:
Dietary Supplement: Vegan diet — Provide

SUMMARY:
The purpose of this study is to evaluate the impact of community health screening, health education and nutritional intervention on risk factors for cardiovascular disease in a predominantly African American population. The health fair and intervention will take place in a church that typically improves their lifestyle by "giving up for Lent" certain foods or habits. Participation in this nutrition intervention is voluntary and each participant will sign an informed consent along with a waiver. On the waiver, the participant can agree to have all testing performed but can withdraw consent at any time or decide to have only some of the testing.

It was hypothesized that a community-based health screening and nutritional intervention will have a positive impact on the participants by:

1. Measuring baseline risk factors
2. Educating them about their individual risk for heart disease
3. Providing education on healthy lifestyle
4. Providing a nutritional intervention for 40 days with home- delivered plant-based meals nutrition that has been shown to lower cardiac risk factors
5. Repeating the risk factor assessment at the end of the intervention, to demonstrate the degree of, if any, reduction in cardiac risk as assessed by the American College of Cardiology/American Heart Association (ACC/AHA) Atherosclerotic Cardiovascular Disease (ASCVD) Risk Calculator
6. Motivating at-risk subjects to seek continued appropriate medical care and to institute more permanent relevant lifestyle changes (e.g., diet, exercise, medication compliance).

DETAILED DESCRIPTION:
Design and Methods:

A prospective study design will be implemented. Approximately 50 participants are expected to volunteer for the intervention. The health screening will consist of measuring stations. After signing an informed consent and a waiver, the participant will complete an intake form, which includes basic patient information and demographics including date of birth, gender, height, and race/ethnicity. Also on the intake form, the participant will list medications currently being taken, risk factors for heart disease (i.e., diabetes, hypertension, hyperlipidemia, and smoking), family history of heart disease, and current medical conditions. After completing the intake form, the participant will have their height, weight, blood pressure, and pulse measured. If the participant uses oxygen regularly or is feeling short of breath, oxygen saturation will be measured using a pulse oximeter. Finally, each participant will have a blood tests for fasting (preferably for 9 hours) blood glucose, hemoglobin A1C, insulin level, lipid profile, high-sensitivity C-reactive protein, small dense LDL cholesterol, lipoprotein a, trimethylamine N-oxide (TMAO) and suPAR at baseline. Each of these parameters will be repeated for comparison at day 40 of Lent (Easter weekend). Blood will be stored for future analysis, since assays for suPAR and TMAO may not be immediately available.

From the information gathered, each participant will be given a baseline American College of Cardiology/American Heart Association (ACC/AHA) Atherosclerotic Cardiovascular Disease (ASCVD) risk score, which is an estimate of the 10-year and lifetime risks of ASCVD (defined as coronary death or nonfatal myocardial infarction, or fatal or nonfatal stroke). After the last visit, health education and counseling will be provided which is tailored to each individual given the findings gathered during the initial screening and the change that occurred. The information gathered will be written down on a form for the participant to keep for his own records. Referrals to primary care physicians, cardiologists, or other healthcare providers will be given as needed after the initial or post-intervention risk assessment. Patients who undergo lipid, blood pressure or glucose lowering therapy between the two assessments will be censured from the appropriate laboratory data analysis.

Subject Selection:

Approximately 50 subjects will be enrolled.

Inclusion Criteria:

1. Age >18
2. Able to consent to dietary protocol
3. Willing to comply with study requirements and voluntarily agrees to participate in this clinical study after appropriate informed consent is provided.

Exclusion Criteria:

1. Vegetarians
2. Inability to regularly measure blood pressure if taking antihypertensive medications
3. Inability to regularly measure blood sugar if taking antihyperglycemic medications
4. Celiac disease (gluten enteropathy)
5. Treatment for eating disorder
6. Active treatment for malignancy
7. Inability to eat solid food
8. Fruit, nut or vegetable allergy

Study Variables:

1. Demographic information (date of birth, race/ethnicity)
2. Height
3. Weight
4. Body mass index (BMI)
5. Patient names, addresses and phone numbers
6. History of known coronary artery disease (CAD)
7. CAD risk factors (age, gender, hypertension, diabetes mellitus (DM), dyslipidemia, current or prior tobacco use, and family history of premature CAD),
8. History of typical angina pectoris,
9. CAD risk equivalents (peripheral or carotid arterial disease, stroke, transient ischemic attack, chronic kidney disease with glomerular filtration rate (GFR) < 60 ml/min/1.7m2 or end-stage renal disease).
10. Medications including aspirin, lipid lowering agent, antihypertensive and antihyperglycemic.
11. Home blood pressure and blood glucose measurements at least 3 days per week.

Laboratory Tests Samples will be collected from individuals being evaluated at the baseline and blood upon re-evaluation at day 40 of Lent:

1. Blood glucose
2. Glycosylated hemoglobin
3. Insulin level
4. Lipid profile
5. High-sensitivity C-reactive protein
6. Small dense low-density lipoprotein (LDL) cholesterol
7. Lipoprotein a
8. trimethylamine oxide (TMAO)
9. soluble urokinase plasminogen activator receptor (suPAR)

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Able to consent to dietary protocol
3. Willing to comply with study requirements and voluntarily agrees to participate in this clinical study after appropriate informed consent is provided.

Exclusion Criteria:

1. Vegetarians
2. Inability to regularly measure blood pressure if taking antihypertensive medications
3. Inability to regularly measure blood sugar if taking antihyperglycemic medications
4. Celiac disease (gluten enteropathy)
5. Treatment for eating disorder
6. Active treatment for malignancy
7. Inability to eat solid food
8. Fruit, nut or vegetable

Inclusion Criteria:

1. Age >18
2. Able to consent to dietary protocol
3. Willing to comply with study requirements and voluntarily agrees to participate in this clinical study after appropriate informed consent is provided.

Exclusion Criteria:

1. Vegetarians
2. Inability to regularly measure blood pressure if taking antihypertensive medications
3. Inability to regularly measure blood sugar if taking antihyperglycemic medications
4. Celiac disease (gluten enteropathy)
5. Treatment for eating disorder
6. Active treatment for malignancy
7. Inability to eat solid food
8. Fruit, nut or vegetable allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
American College of Cardiology/American Heart Association (ACC/AHA) Atherosclerotic Cardiovascular Disease (ASCVD) Risk Calculator, ranging from 1% to 50% 10-year event risk | 5 weeks
  ACC/AHA Guideline for Prevention Tool calculated based on blood pressure, total cholesterol, HDL cholesterol, diabetes, age, gender, ethnicity, and smoking history.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No